CLINICAL TRIAL: NCT04357340
Title: Efficacy of Pulmonary Physiotherapy on Hospitalized Patients With Novel Coronavirus 2019 Pneumonia
Brief Title: The Effects of Pulmonary Physiotherapy Treatments on Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Javaherian, PhD. Candidate of Phyiotherapy, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99-1-103-47429
Record Dates: First submitted 2020-04-13; First posted 2020-04-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; Pneumonia; SARS Pneumonia
Keywords: Pulmonary Physiotherapy; 2019 novel coronavirus disease; COVID-19; Rehabilitation
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: All the enrolled participants will be allocated to the intervention of control groups using blocked-balanced randomization method.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Physiotherapy Techniques group (Experimental): Pulmonary physiotherapy techniques, 6 sessions during 3 days and incentive spirometer.
  Interventions: Other: Pulmonary Physiotherapy Techniques
- Control group (No Intervention): Incentive spirometer only

INTERVENTIONS:
Other: Pulmonary Physiotherapy Techniques — Participants will receive pulmonary physiotherapy techniques in six session during three days (twice daily). Four distinguished interventions will be provided for the patients: 1) Chest expansion exercises (for prevention and treatment of potential atelectasis); 2) Techniques to Mobilize or loosen the pulmonary secretions (Active cycle breathing, Coughing techniques, Vibration and Postural drainage); 3) Hold breathing exercise (3 sets, 10 repetition) and; 4) Walking training (based on patient's tolerance until 6 minute).
  Arms: Pulmonary Physiotherapy Techniques group

SUMMARY:
The aim of this study is to evaluate the efficacy of pulmonary physiotherapy on respiratory functions in hospitalized patients with Novel Coronavirus 2019 pneumonia. Patients will be randomized into 1) intervention group: receiving pulmonary physiotherapy technique to improve pulmonary function and walking training or 2) control group: Usual medical care. Patients in both groups will receive therapeutic incentive spirometer. Various outcome measurements of pulmonary functions will be evaluated before and after of interventions. Mortality rate, hospitalization duration and re-admission will be followed until one month after end of intervention. Also, patient's quality of life will be measured after one month.

DETAILED DESCRIPTION:
In late December 2019, the new coronavirus (COVID-19) emerged in Wuhan, China and it has been confirmed as the cause of pneumonia in a large number of Chinese patients. The virus, also known as SARS-CoV-2, has since then spread to more than 200 countries worldwide.

The most common symptoms of COVID-19 are fever, dry cough, shortness of breath and tiredness. In severe cases, the infection could cause pneumonia, acute respiratory distress syndrome (ARDS) and sometimes leads to death. Pulmonary physiotherapy is a comprehensive, effective and safe treatment method which is aimed at improving patient's respiratory symptoms, train effective coughing, clear the airway secretion, eliminate exacerbation and so on. It seems that pulmonary physiotherapy interventions can effectively decrease hospitalization, reduce the risk of complications and improve the patient's medical condition.

The aim of this study is to evaluate the effectiveness of the hold breathing technique, chest expansion exercise, postural drainage procedure and Cough techniques carried out during pulmonary physiotherapy sessions.

The researchers will invite 40 hospitalized patients in Imam Khomeini Hospital Complex, Tehran, Iran. All patients will be enrolled after taking informed consent. All of the procedure will be performed with the coordination of the patient's physicians. Patients will be randomized to the intervention or control group. Primary outcome measurements will be evaluated immediately before and after the interventions (with three days period). Also, patient's condition (including process of disease progression, mortality, hospital stay duration and re-admission) will be followed until one month using medical records review and interviewing with the patient or his/her family. Patient's health related quality of life will be measured using short form-36 quality of life assessment tool one month after the end of interventions. Intention-to-treat analysis will be performed in the patients that dropped out of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with COVID-19 pneumonia confirmed by RT-PCR test and diagnostic radiology.
2. Non-intubated patients
3. Patients with full consciousness
4. Be able to walking and performing exercises.
5. O2 Saturation < 88% when free air breathing.
6. be able to write and read in Farsi

Exclusion Criteria:

1. Any type of musculoskeletal disorder disabling patient to participate to study.
2. Intubation during the period of intervention
3. Patients' dissatisfaction to continue the study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Mixed venous O2 pressure (PVO2) | Baseline
  Partial pressure of oxygen in mixed venous blood.
Mixed venous O2 pressure (PVO2) | Day 3
  Partial pressure of oxygen in mixed venous blood.
Mixed venous CO2 pressure (PVCO2) | Baseline
  Partial pressure of carbon dioxide in mixed venous blood.
Mixed venous CO2 pressure (PVCO2) | Day 3
  Partial pressure of carbon dioxide in mixed venous blood.
PH | Baseline
  Measure of the venous blood acidity or alkalinity
PH | Day 3
  Measure of the venous blood acidity or alkalinity
HCO3 | Baseline
  The amount of bicarbonate ion in the venous blood
HCO3 | Day 3
  The amount of bicarbonate ion in the venous blood
Oxygen saturation (O2 Sat) from VBG | Baseline
  The amount of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the venous blood
Oxygen saturation (O2 Sat) from VBG | Day 3
  The amount of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the venous blood
Three minute walk test | Baseline
  The distance a patient can walk during three minute
Three minute walk test | Day 3
  The distance a patient can walk during three minute
O2 Sat after one minute walking | Baseline
O2 Sat after one minute walking | Day 3
O2 Sat after two minutes use of Partial Rebreather | Baseline
O2 Sat after two minutes use of Partial Rebreather | Day 3
O2 Sat after two minutes free air breathing | Baseline
O2 Sat after two minutes free air breathing | Day 3
O2 sat/ Fio2 | Baseline
O2 sat/ Fio2 | Day 3

SECONDARY OUTCOMES:
Mortality rate | until one month
  The number of dead subjects compared to total patients
Number of participants with Rehospitalization | until one moth
  Patients' hospitalization after discharge due to any reason
The Health-Related Quality of Life (HRQOL) | One month after end of intervention
  Using Short-form 36 questionnaire. The minimum score is 0 and the maximum score is 100. Higher scores mean patient's better quality of life.
breathlessness | Baseline
  The amount of shortness of breath using Visual Analogue Scale (VAS). The minimum score is 0 and maximum is 10. The 0 score means no breathlessness and the 10 score is the maximum breathlessness.
breathlessness | Day 3
  The amount of shortness of breath using Visual Analogue Scale (VAS). The minimum score is 0 and maximum is 10. The 0 score means no breathlessness and the 10 score is the maximum breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Javaherian, Ph.D. cand., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital Complex, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after de-identification
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 12 months following article publication
Access Criteria: Researchers who provide an approved methodologically proposal in the same purpose

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Read JM, Bridgen JRE, Cummings DAT, Ho A, Jewell CP. Novel coronavirus 2019-nCoV (COVID-19): early estimation of epidemiological parameters and epidemic size estimates. Philos Trans R Soc Lond B Biol Sci. 2021 Jul 19;376(1829):20200265. doi: 10.1098/rstb.2020.0265. Epub 2021 May 31. PMID 34053269
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chen J. Pathogenicity and transmissibility of 2019-nCoV-A quick overview and comparison with other emerging viruses. Microbes Infect. 2020 Mar;22(2):69-71. doi: 10.1016/j.micinf.2020.01.004. Epub 2020 Feb 4. PMID 32032682
- [Background] Liu T, Hu J, Kang M, Lin L, Zhong H, Xiao J, et al. Transmission dynamics of 2019 novel coronavirus (2019-nCoV). 2020.
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Bott J, Blumenthal S, Buxton M, Ellum S, Falconer C, Garrod R, Harvey A, Hughes T, Lincoln M, Mikelsons C, Potter C, Pryor J, Rimington L, Sinfield F, Thompson C, Vaughn P, White J; British Thoracic Society Physiotherapy Guideline Development Group. Guidelines for the physiotherapy management of the adult, medical, spontaneously breathing patient. Thorax. 2009 May;64 Suppl 1:i1-51. doi: 10.1136/thx.2008.110726. No abstract available. PMID 19406863
- [Background] Strickland SL, Rubin BK, Haas CF, Volsko TA, Drescher GS, O'Malley CA. AARC Clinical Practice Guideline: Effectiveness of Pharmacologic Airway Clearance Therapies in Hospitalized Patients. Respir Care. 2015 Jul;60(7):1071-7. doi: 10.4187/respcare.04165. PMID 26113566
- [Background] Yang F, Liu N, Hu JY, Wu LL, Su GS, Zhong NS, Zheng ZG. [Pulmonary rehabilitation guidelines in the principle of 4S for patients infected with 2019 novel coronavirus (2019-nCoV)]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):180-182. doi: 10.3760/cma.j.issn.1001-0939.2020.03.007. Chinese. PMID 32164083
- [Background] Jin X, Lian JS, Hu JH, Gao J, Zheng L, Zhang YM, Hao SR, Jia HY, Cai H, Zhang XL, Yu GD, Xu KJ, Wang XY, Gu JQ, Zhang SY, Ye CY, Jin CL, Lu YF, Yu X, Yu XP, Huang JR, Xu KL, Ni Q, Yu CB, Zhu B, Li YT, Liu J, Zhao H, Zhang X, Yu L, Guo YZ, Su JW, Tao JJ, Lang GJ, Wu XX, Wu WR, Qv TT, Xiang DR, Yi P, Shi D, Chen Y, Ren Y, Qiu YQ, Li LJ, Sheng J, Yang Y. Epidemiological, clinical and virological characteristics of 74 cases of coronavirus-infected disease 2019 (COVID-19) with gastrointestinal symptoms. Gut. 2020 Jun;69(6):1002-1009. doi: 10.1136/gutjnl-2020-320926. Epub 2020 Mar 24. PMID 32213556
- [Background] Novoa N, Ballesteros E, Jimenez MF, Aranda JL, Varela G. Chest physiotherapy revisited: evaluation of its influence on the pulmonary morbidity after pulmonary resection. Eur J Cardiothorac Surg. 2011 Jul;40(1):130-4. doi: 10.1016/j.ejcts.2010.11.028. Epub 2011 Jan 11. PMID 21227711
- [Background] Ambrosino N, Makhabah DN. Comprehensive physiotherapy management in ARDS. Minerva Anestesiol. 2013 May;79(5):554-63. Epub 2013 Jan 10. PMID 23306398
- [Background] Munshi L, Kobayashi T, DeBacker J, Doobay R, Telesnicki T, Lo V, Cote N, Cypel M, Keshavjee S, Ferguson ND, Fan E. Intensive Care Physiotherapy during Extracorporeal Membrane Oxygenation for Acute Respiratory Distress Syndrome. Ann Am Thorac Soc. 2017 Feb;14(2):246-253. doi: 10.1513/AnnalsATS.201606-484OC. PMID 27898220
- [Background] Paulus F, Binnekade JM, Vroom MB, Schultz MJ. Benefits and risks of manual hyperinflation in intubated and mechanically ventilated intensive care unit patients: a systematic review. Crit Care. 2012 Aug 3;16(4):R145. doi: 10.1186/cc11457. PMID 22863373
- [Background] Hillegass E. Essentials of Cardiopulmonary Physical Therapy-E-Book: Elsevier Health Sciences; 2016.
- [Background] Iriberri M, Galdiz JB, Gorostiza A, Ansola P, Jaca C. Comparison of the distances covered during 3 and 6 min walking test. Respir Med. 2002 Oct;96(10):812-6. doi: 10.1053/rmed.2002.1363. PMID 12412981
- [Background] Pan AM, Stiell IG, Clement CM, Acheson J, Aaron SD. Feasibility of a structured 3-minute walk test as a clinical decision tool for patients presenting to the emergency department with acute dyspnoea. Emerg Med J. 2009 Apr;26(4):278-82. doi: 10.1136/emj.2008.059774. PMID 19307390
- [Derived] Javaherian M, Shadmehr A, Keshtkar A, Beigmohammadi MT, Dabbaghipour N, Syed A, Attarbashi Moghadam B. Safety and efficacy of pulmonary physiotherapy in hospitalized patients with severe COVID-19 pneumonia (PPTCOVID study): A prospective, randomised, single-blind, controlled trial. PLoS One. 2023 Jan 31;18(1):e0268428. doi: 10.1371/journal.pone.0268428. eCollection 2023. PMID 36719885